CLINICAL TRIAL: NCT00003798
Title: Phase I Study Involving Gadolinium Texaphyrin (NSC 695238) in Patients With Pancreatic and Periampullary Adenocarcinoma Receiving Radiotherapy for Unresectable Disease
Brief Title: Radiation Therapy Plus Gadolinium Texaphyrin in Treating Patients With Cancer of the Pancreas That Cannot Be Removed by Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: CDR0000066941, J9840; P30CA006973 (NIH); JHOC-98062407; NCI-T97-0115
Record Dates: First submitted 1999-11-01; First posted 2004-08-04 (Estimated); Last update posted 2012-11-14 (Estimated); Status verified 2012-11

CONDITIONS: Pancreatic Cancer
Keywords: stage II pancreatic cancer; stage III pancreatic cancer; adenocarcinoma of the pancreas
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — motexafin gadolinium; Radiotherapy

INTERVENTIONS:
Drug: motexafin gadolinium
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to damage tumor cells. Drugs such as gadolinium texaphyrin may make the tumor cells more sensitive to radiation therapy.

PURPOSE: Phase I trial to study the effectiveness of gadolinium texaphyrin plus radiation therapy in treating patients who have cancer of the pancreas that cannot be removed by surgery.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose of gadolinium texaphyrin in patients with locally advanced, unresectable pancreatic or periampullary adenocarcinoma undergoing local regional radiotherapy. II. Determine the toxic effects of gadolinium texaphyrin with concurrent radiotherapy in these patients. III. Correlate estimates of tumor and normal organ gadolinium texaphyrin uptake and retention over time by MRI with plasma/serum levels in these patients.

OUTLINE: This is a dose escalation study. Patients receive gadolinium texaphyrin IV over 5-10 minutes 4 times weekly at least 2 hours prior to external beam radiotherapy over 2.5 weeks (total of 10 fractions). Cohorts of 3-6 patients are treated at escalating doses of gadolinium texaphyrin. The maximum tolerated dose is defined as the highest dose level in which dose limiting toxicity occurs in no more than 2 of 6 patients. Patients are followed once monthly for 2 months.

PROJECTED ACCRUAL: A total of 45 evaluable patients will be accrued for this study within 18-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed locally advanced, unresectable pancreatic or periampullary adenocarcinoma Patients may have evidence of hepatic or other intra-abdominal or systemic metastases if they have dominant symptomatology from the locally unresectable component of disease Prior treatment with 1 chemotherapy regimen required Palliative bypass procedures without resection allowed Bidimensionally measurable disease on CT or MRI scan

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: Karnofsky 60-100% Life expectancy: Not specified Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 150,000/mm3 Hemoglobin at least 8.5 g/dL No history of G6PD deficiency Hepatic: SGOT or SGPT less than 2 times upper limit of normal (ULN) Alkaline phosphatase less than 2 times ULN Bilirubin no greater than 2.0 mg/dL (elevated values must be falling or stable for at least 1 week prior to therapy) Renal: Creatinine no greater than 2.0 mg/dL (no clinical indication of compromised kidney) Other: Not pregnant or nursing Fertile patients must use effective contraception No second malignancy within the past 5 years, except: Resected superficial nonmelanomatous skin cancer Carcinoma in situ of the cervix No uncontrolled or serious medical conditions No active peptic ulcers No weight loss greater than 5% of ideal body weight within 30 days prior to study No uncontrolled nausea and vomiting No claustrophobia

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 4 weeks since prior biologic therapy No concurrent experimental biologic therapy Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: No prior radiotherapy compromising the delivery of radiation on this study No prior radiotherapy to areas within the planned field of treatment Surgery: At least 4 weeks since prior gastrointestinal surgery Other: At least 4 weeks since prior experimental drugs No other concurrent experimental drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2000-04

CONTACTS AND LOCATIONS:
Overall Officials: Ross A. Abrams, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (1):
- Johns Hopkins Oncology Center, Baltimore, Maryland, United States